CLINICAL TRIAL: NCT02364063
Title: Micturition Reeducation in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/766.1
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Daytime Urinary Incontinence
Keywords: Urinary incontinence; cerebral palsy; urotherapy; child
MeSH Terms: conditions — Diurnal Enuresis; Urinary Incontinence; Cerebral Palsy | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Children with CP - Therapy (Experimental): Children receive incontinence treatment during one year, after which a follow-up period of 6 months will be applied. Intervention includes standard urotherapy with or without pharmacotherapy/specific urotherapy
  Interventions: Other: urotherapy with or without pharmacotherapy
- Children with CP - Control (No Intervention): Children are followed for 6 months, not receiving any treatment. After this follow-up period, children also receive incontinence treatment for 6 months.
- Children without CP (Active Comparator): Children receive incontinence treatment during 1 year. Intervention includes standard urotherapy with or without pharmacotherapy/specific urotherapy
  Interventions: Other: urotherapy with or without pharmacotherapy

INTERVENTIONS:
Other: urotherapy with or without pharmacotherapy — Individualized
  Arms: Children with CP - Therapy; Children without CP

SUMMARY:
This study evaluates the effectiveness of a voiding reeducation program as treatment for incontinence in children with a brain injury.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) (Rosenbaum, 2007) gain bladder and bowel control at older age compared to typical developing children (Ozturk, 2006). The incidence of urinary incontinence during day and night, fecal incontinence and constipation is higher in this population.

Incontinence in children is often treated with urotherapy. This is a nonsurgical, nonpharmacological treatment for lower urinary tract dysfunctions. Standard urotherapy is noninterventional and it includes giving information, instructions, advice regarding life-style, fluid intake and bladder diaries. Additionally specific interventions can be used, such as: various forms of pelvic floor training, behavioral modification, biofeedback, electrical stimulation and catheterization (Neveus, 2006). Recent research has proven urotherapy to be successful for the treatment of children with daytime incontinence (Mulders, 2010).

Despite the high prevalence of incontinence in children with CP the possible treatment strategies in this population are poorly investigated. Far too often, urinary incontinence in children with CP is considered a normal, unavoidable and even a minor problem.

Aim: Investigate the influence of individualized urotherapy on the (in)continence of children with CP.

The included children with CP will be randomized and stratified for type of CP and mental abilities into 2 groups: the intervention group and the control group. The intervention group will receive immediate therapy. After one year of therapy, a follow- up of 6 months will be applied. The control group will start 6 months later and information will be used as control group. Incontinent children without CP will receive therapy and will also act as control group.

ELIGIBILITY:
Inclusion Criteria:

* Daytime urinary incontinence with or without enuresis and/or fecal incontinence
* Cerebral palsy (Arms of children with CP)
* Normal development (Arms of children without CP)

Exclusion Criteria:

* Isolated urinary tract infections
* Isolated enuresis
* Isolated dysfunctional voiding
* Isolated fecal incontinence
* Anatomical abnormalities
* History of genitourinary or renal surgery
* Medication for incontinence during the last 3 months
* Pelvic reeducation during the last 6 months
* other neurologic problems influencing continence

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Subjective report of change in urinary incontinence measured by questionnaire | Baseline and 3-6-12 months + follow-up

SECONDARY OUTCOMES:
Lower urinary tract symptoms (LUTS) measured by questionnaire | baseline and 6-12 months
Drinking behaviour measured by drinking and voiding charts | Baseline and 6-12 months
Constipation/fecal incontinence measured by ROME III criteria | Baseline and 6-12 months
voiding variables and pelvic floor activity during micturition measured by uroflow/EMG | Baseline and 3-6-12 months
  Uroflow and pelvic floor EMG + postmictional residue

CONTACTS AND LOCATIONS:
Overall Officials: Erik Van Laecke, PhD MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Samijn B, Van den Broeck C, Plasschaert F, Pascal A, Deschepper E, Hoebeke P, Van Laecke E. Incontinence training in children with cerebral palsy: A prospective controlled trial. J Pediatr Urol. 2022 Aug;18(4):447.e1-447.e9. doi: 10.1016/j.jpurol.2022.05.014. Epub 2022 May 25. PMID 35732572